CLINICAL TRIAL: NCT01580358
Title: Changhua Christian Hospital
Brief Title: Therapeutic Effects of Traditional Chinese Medicine, Shen-Mai San in Cancer Patient Undergoing Chemotherapy or Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhua Christian Hospital (Other)
Collaborators: Committee on Chinese Medicine and Pharmacy (Other Government)
Responsible Party: Principal Investigator, Chia-Yun Chen, MD, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CCMP98 -CT-203
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Cancer Patients Undergoing Chemotherapy or Radiotherapy
Keywords: cancer; radiotherapy; chemotherapy; Traditional Chinese Medicine; Safety
MeSH Terms: conditions — Neoplasms | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shen-Mai San (Active Comparator): Shen mai san is composed of three herb medicines, Ginseng radis, Liriope spicata, and Schizandrae fructus and was manufactured into concentrated herbal extract and packed with 0.5g per capsule and labeled by Sun-Ten pharmaceutical company in Taiwan with good manufacturing practice (GMP).
  Interventions: Drug: Shen-Mai San
- starch (Placebo Comparator): Starch in the same granule as intervention group for this double-blind trial
  Interventions: Drug: Starch

INTERVENTIONS:
Drug: Shen-Mai San — Shen mai san is composed of three herb medicines, Ginseng radis, Liriope spicata, and Schizandrae fructus and was manufactured into concentrated herbal extract and packed with 0.5g per capsule and labeled by Sun-Ten pharmaceutical company in Taiwan with good manufacturing practice (GMP).
  Arms: Shen-Mai San
Drug: Starch — It was packed in granules with 0.5gm starch. Patients took eight granules three times per day for four weeks.
  Arms: starch

SUMMARY:
Using Shen-Mai-San for cancer patients undergoing chemotherapy or radiotherapy could help these people improve the quality of life.

DETAILED DESCRIPTION:
Shen-Mai-San could improve fatigue, general weakness, neutropenia for patients under going chemotherapy or radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative patients with histologically confirmed cancer within 3 years and undergoing chemotherapy or radiotherapy
* age above 18 years old
* signed informed consent
* ability to read Chinese, ability for oral intake.

Exclusion Criteria:

* being pregnancy
* on breast feeding
* completed chemotherapy or radiotherapy
* brain metastasis with Eastern Cooperative Oncology Group (ECOG) performance status of two to four
* delusion or hallucination
* acute infection
* received medications for other clinical trials.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in EORTC QOL-C30 at four weeks | baseline and four weeks

SECONDARY OUTCOMES:
Change from baseline in BUN, Creatinine, GOT, GPT at four weeks | baseline and four weeks
  monitor the liver function and renal function
Change from baseline in Heart rate variability at four weeks | baseline and four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lun Chien Lo, MD. PhD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

REFERENCES:
- [Derived] Lo LC, Chen CY, Chen ST, Chen HC, Lee TC, Chang CS. Therapeutic efficacy of traditional Chinese medicine, Shen-Mai San, in cancer patients undergoing chemotherapy or radiotherapy: study protocol for a randomized, double-blind, placebo-controlled trial. Trials. 2012 Dec 3;13:232. doi: 10.1186/1745-6215-13-232. PMID 23206440